CLINICAL TRIAL: NCT01838720
Title: Zero Ischemia Laparoscopic Radio Frequency Ablation Assisted Enucleation of Renal Cell Carcinoma With T1a Stage : Clinical Outcomes of a Randomised Controlled Trial
Brief Title: Zero Ischemia Laparoscopic Radio Frequency Ablation Assisted Enucleation of Renal Cell Carcinoma With T1a Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yiran Huang, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-20130406
Record Dates: First submitted 2013-04-14; First posted 2013-04-24 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Renal Cell Carcinoma; Zero Ischemia
Keywords: renal cell carcinoma; ischemia; radio frequency ablation
MeSH Terms: conditions — Carcinoma, Renal Cell; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zero ischemia laparoscopic RFA assisted TE (Experimental): RFA will be performed for 1 to 4 cycles for 4 to 12 minutes each depending on tumor size and depth. The tumor then will be laparoscopic enucleation without hilar clamping.
  Interventions: Procedure: zero ischemia laparoscopic RFA assisted TE
- conventional laparoscopic partial nephrectomy (Active Comparator): Renal hilum will be accurately isolated and then the artery only will be clamped during surgery.
  Interventions: Procedure: ischemia

INTERVENTIONS:
Procedure: zero ischemia laparoscopic RFA assisted TE
  Other Names: zero ischemia laparoscopic radio frequency ablation assisted tumor enucleation
  Arms: zero ischemia laparoscopic RFA assisted TE
Procedure: ischemia — conventional laparoscopic partial nephrectomy
  Other Names: renal artery will be clamped during surgery.
  Arms: conventional laparoscopic partial nephrectomy

SUMMARY:
To evaluate the feasibility and efﬁciency of zero ischemia laparoscopic radio frequency ablation assisted enucleation of T1a renal cell carcinoma in comparison with the conventional laparoscopic partial nephrectomy.

DETAILED DESCRIPTION:
Warm ischemic injury is one of the most important factors affecting renal function in partial nephrectomy (PN). Zero ischemia partial nephrectomy technique using renal arterial branch microdissection could protect renal function during surgery, but it requires longer operative time and more blood loss than conventional partial nephrectomy. The technique of zero ischemia laparoscopic radio frequency ablation assisted enucleation of renal cell carcinoma appears to be an alternative that eliminates warm ischemia, preserves the maximal parenchyma and is oncologically safe. Our study was designed to evaluate this technique in comparison with the conventional laparoscopic partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with sporadic, unilateral, newly diagnosed T1a presumed renal cell carcinoma
* patients with normal contralateral renal function (diﬀerential renal function of >40% as determined by radionuclide scintigraphy)
* patients agreeable to participate in this long-term follow-up study

Exclusion Criteria:

* patients' aged >80 years
* patients with other renal diseases
* patients not able to tolerate the laparoscopic procedure
* patients with previous renal surgery or history of any inﬂammatory conditions of the operative kidney
* patients with the renal tumor close to the calyces

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
the absolute change in glomerular ﬁltration rate (GFR) of the aﬀected kidney | baseline and 12 months
  12 months minus baseline

SECONDARY OUTCOMES:
estimated GFR (eGFR) | 12 months
changes in GFR of total kidneys by renal scintigraphyby | baseline and 12 months
blood loss | during surgery
surgical margin | postoperative
  pathologic confirm of surgical margin
postoperative complications | 12 months
progression-free survival | 12 months
local recurrence | 12 months
the absolute change in glomerular ﬁltration rate (GFR) of the aﬀected kidney | baseline and 6 months
  6 months minus baseline
estimated GFR (eGFR) of 6 month | 6 month
changes in GFR of total kidneys by renal scintigraphyby of 6 month | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Yiran Huang, M.D., Principal Investigator — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang J, Zhang J, Wang Y, Kong W, Xue W, Liu D, Chen Y, Huang Y. Comparing Zero Ischemia Laparoscopic Radio Frequency Ablation Assisted Tumor Enucleation and Laparoscopic Partial Nephrectomy for Clinical T1a Renal Tumor: A Randomized Clinical Trial. J Urol. 2016 Jun;195(6):1677-83. doi: 10.1016/j.juro.2015.12.115. Epub 2016 Feb 22. PMID 26905020